CLINICAL TRIAL: NCT06589791
Title: A Disease Area Study on the Awareness and Perceptions of Systemic Inflammation and hsCRP as a biomARKer in Patients With ASCVD and CKD in China Among Cardiologists and Nephrologists
Acronym: SPARK-CVD
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: DAS-8091; U1111-1303-3098 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Atherosclerotic Cardiovascular Disease (ASCVD); Chronic Kidney Disease (CKD)
MeSH Terms: conditions — Atherosclerosis; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Health care professionals: Cardiologists and nephrologists in China
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — Online self-completion survey

SUMMARY:
This is a survey-based study with the objective to understand the awareness, perceptions and potential clinical management patterns among Chinese cardiologists and nephrologists towards the role of systemic inflammation in patients with ASCVD and CKD in real-world clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Work in cardiology, internal medicine, or nephrology department
* Specialize in one of the following: coronary interventional cardiology, HF, general cardiology, preventive cardiology, cardiac rehabilitation or nephrology
* Practice at consultant level for 3+ years after standardized training for resident physicians or 3+ years' working experience as a specialist
* Manage at least 20 adult patients with ASCVD and CKD (not dialysis-only) every month

Exclusion Criteria:

* Unwilling to provide informed consent
* Insufficient number of patients with ASCVD and CKD
* Do not fulfil inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiologists and nephrologists with patients that have ASCVD and CKD in China
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Health care professional's perceptions towards the role of systemic inflammation in the identification, treatment and management of patients with ASCVD and CKD | At the time of survey response (Day 1)
  Multi-select from a defined list; Single-select from a defined list; Numerical; 7-point Likert scale for measurement of agreement to different statements from 1 "strongly disagree" to 7 "strongly agree"

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Shanghai Pharmaceuticals Co., Ltd, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com